CLINICAL TRIAL: NCT00981955
Title: A Randomised, Double Blind, Placebo-controlled Study to Evaluate the Effects of Caffeine and L-theanine Both Alone and in Combination on Cerebral Blood Flow, Cognition and Mood.
Brief Title: The Effects of Caffeine and L-theanine Both Alone and in Combination on Cerebral Blood Flow, Cognition and Mood
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Dr Crystal Haskell, Northumbria University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 25AA1
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2010-07

CONDITIONS: Cognitive Function; Mood
Keywords: Caffeine; Ltheanine; Near Infrared Spectroscopy; Cerebral Blood Flow; Cognitive Function; Mood
MeSH Terms: interventions — Caffeine; theanine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 75mg caffeine (Active Comparator)
  Interventions: Dietary Supplement: Caffeine and L-theanine
- 50mg l-theanine (Active Comparator)
  Interventions: Dietary Supplement: Caffeine and L-theanine
- 75mg caffeine and 50mg l-theanine (Active Comparator)
  Interventions: Dietary Supplement: Caffeine and L-theanine
- 0mg caffeine/l-theanine (Placebo Comparator)
  Interventions: Dietary Supplement: Caffeine and L-theanine

INTERVENTIONS:
Dietary Supplement: Caffeine and L-theanine — Acute oral administration of 75mg of caffeine, 50mg l-theanine, 75mg caffeine and 50mg l-theanine in combination or placebo. One dosage administered on each of four separate study days.
  Other Names: Sun-theanine (l-theanine)

SUMMARY:
Although the beneficial effects of caffeine on cognition and mood have been reported in a number of studies, relatively few studies have looked at the effects of caffeine in combination with other phytonutrients despite the fact that caffeine is seldom consumed in isolation. L-theanine is a naturally occurring amino-acid found in tea, and has been used historically as a relaxing agent (Haskell et al., 2008). Few have assessed the impact of l-theanine on cognition, but of those that have, the most interesting results were obtained when l-theanine was assessed in combination with caffeine (Haskell et al., 2008). It remains unclear what is underlying the reported effects.

Near Infrared Spectroscopy (NIRS) is an emerging neuroimaging technology that is capable of determining changes in cerebral blood flow (CBF) by measuring the optical properties of oxygenated and deoxygenated blood (Bunce et al., 2006). No study to date has used NIRS to assess cerebral blood flow following treatment with either caffeine, l-theanine or a combination of both. It is anticipated that the proposed study will provide some insight into the mechanism of the previously observed effects both alone and in combination.

A randomised, double-blind, placebo controlled, balanced crossover design study will assess the effects of 75mg caffeine, 50mg l-theanine and a 75mg caffeine/50mg l-theanine combination in 24 young healthy adults (18-35). Cognitive and mood assessments will take place at baseline and at 30 minutes following treatment whilst cerebral haemodynamics are measured via the technique of NIRS.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Aged 18-35
* Either caffeine consumers (consume more than 150mg caffeine per day) or non-consumers (less than 44mg caffeine per day).

Exclusion Criteria:

* Smoke or consume any tobacco products
* Not proficient in English language
* Pregnant (or seeking to become pregnant)
* Taking recreational, over the counter/prescription medication (including the contraceptive pill), and/or dietary/herbal supplements
* Have food allergies or sensitivities
* Have history of/current head trauma, learning difficulties , ADHD, migraines or any gastric problems

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-08; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Cerebral blood flow | 0-80 minutes post dose
Cognitive function | 0-70 minutes post-dose
Mood | 85 minutes post dose

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Haskell, PhD, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne & Wear, United Kingdom